CLINICAL TRIAL: NCT02321566
Title: Motor Cortex Stimulation for the Treatment of Chronic Facial, Upper Extremity, and Throat Pain.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Device manufacturer no longer supports implant covered under the IDE.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NA_00093333
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Trigeminal Neuralgia (Burchiel Type I); Trigeminal Neuralgia (Burchiel Type II); Trigeminal Neuropathic Pain; Trigeminal Deafferentation Pain; Complex Regional Pain Syndrome (Types I and II, Involving the Upper Extremity); Glossopharyngeal Neuralgia; Upper Extremity Pain Due to Deafferentation of the Cervical Spine; Central Pain Syndromes
MeSH Terms: conditions — Trigeminal Neuralgia; Complex Regional Pain Syndromes; Glossopharyngeal Nerve Diseases

ARMS (1):
- Treatment Arm (Experimental): A craniotomy will be performed for the placement of an epidural motor cortex stimulation lead in the context of subjects with chronic facial, upper extremity, and throat pain. If the stimulation is successful during a trial period with externalized lead cabling, the system cabling will be internalized and connected to an internal implantable pulse generator to power and control the system for the duration of the trial.
  Interventions: Device: Epidural Motor Cortex Stimulation

INTERVENTIONS:
Device: Epidural Motor Cortex Stimulation

SUMMARY:
This study is an open-label study to determine the feasibility of Motor Cortex Stimulation (MCS) in the treatment of patients with chronic pain of the face or upper extremity. MCS will be delivered by use of an electrode and pulse generator, which are FDA approved for spinal cord stimulation but are not approved for MCS. The study has as a single-arm design with the subject at baseline serving as a control for the response to MCS.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females who are greater than 18 years of age.
2. Subject has a diagnosis of chronic pain involving the face, upper extremity, or throat, as determined by a review of medical records, history and physical examination. The types of chronic pain eligible for the study are:

   1. Facial pain, including trigeminal neuralgia Type 1, trigeminal neuralgia Type 2, trigeminal neuropathic pain, trigeminal deafferentation pain, symptomatic trigeminal neuralgia, and postherpetic neuralgia.
   2. Complex Regional Pain Syndrome (Types I and II) involving the arm.
   3. Both chronic and episodic forms of refractory Glossopharyngeal Neuralgia (GN).
   4. Deafferentation of the cervical spine leading to pain of the upper extremity.
   5. Central pain syndromes resulting from a prior cerebrovascular insult occurring at least 5 years prior to the study.
3. Subject determined to be treatment-resistant for at least one year prior to the Screening Visit as demonstrated by clinical evidence (determined by review of medical records and discussion with referring pain specialist, anesthesiologist, or neurologist treating chronic pain). The patient must not have responded to treatment with three adequate regimens of medication including one in each of the following categories: antiepileptic drugs, opioids, and antidepressant medications. The trial period for each medication should be at least four weeks, and the two trials must be within the previous 5 years.
4. Subject has at least a score of 6 on the Visual Analog Scale of Pain at all three clinic visits prior to undergoing surgery.
5. Subject must be ambulatory.
6. Females who are postmenopausal, physically incapable of childbearing, or practicing an acceptable method of birth control. Acceptable methods of birth control include surgical sterilization, hormonal contraceptives, or double-barrier methods (condom or diaphragm with a spermicidal agent or intrauterine device [IUD]). If practicing an acceptable method of birth control, a negative urine pregnancy test result has been obtained at baseline Visits 1 and 2.
7. Subject is assessed by psychologist with respect to i) the role of psychological factors, including psychological comorbidities, in their chronic pain, ii) their ability to rate pain and make decisions during the extraoperative stimulation trial, and iii) to participate in decision-making capacity to provide informed consent.
8. Subject is able to read English, understand and cooperate with study procedures, and has signed a written informed consent form prior to any study procedures.

Exclusion Criteria:

1. Subject had major surgery within three months prior to Baseline Visit 1 or has other surgery planned during the proposed study period.
2. Subject is determined by medical consultant to have medical contraindications to undergoing surgery.
3. Subject is pregnant or breast-feeding.
4. Subject has a history of alcohol or drug abuse within the past 6 months and dependence within the past year.
5. Subject has a medical illness/condition, co-morbid psychiatric illness, and/or abnormal diagnostic finding that would interfere with the completion of the study, confound the results of the study, or pose risk to the patient.
6. Subject has a diagnosis of mental retardation.
7. Subject has a distinct neurological condition not included in the list of chronic pain syndromes studied in this protocol, or a history of traumatic brain injury associated with loss of consciousness of > 1 hour and/or intracranial/epidural/subdural bleeding.
8. Diagnosis of a somatoform pain disorder.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-02; Primary Completion 2017-11-21 (Actual); Study Completion 2017-11-21 (Actual)

PRIMARY OUTCOMES:
Pain Assessments | 58 weeks after trial entry
  As measured by the VAS scale of Pain Intensity and Unpleasantness, the McGill Pain questionnaire, and the Leeds Assessment of Neuropathic Signs and Symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Frederick A Lenz, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- The Johns Hopkins Hospital, Baltimore, Maryland, United States